CLINICAL TRIAL: NCT05367726
Title: The Contributions of the Multidisciplinary Management of TKA Infections in a Reference Center: A Retrospective Study About 52 Cases.
Brief Title: The Contributions of the Multidisciplinary Management of Prosthesis Knee Infections in a Reference Center: A Retrospective Study About 52 Cases.Skin Coverage in a Reference Center: A Retrospective Study About 52 Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 776
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Knee Joint Prosthesis Infection; Flap Necrosis; Skin Graft Complications
Keywords: knee joint prosthesis; Flap; Skin Graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having had skin coverage of the knee: patients having had skin coverage of the knee after or at the same time than an orthopedic surgery to treat a knee prosthesis infection
  Interventions: Other: patients having had skin coverage of the knee

INTERVENTIONS:
Other: patients having had skin coverage of the knee — the cutaneous cover is not always optimal to protect the prosthesis, an act of reconstructive plastic surgery is then necessary

SUMMARY:
Acute and chronic infection of knee joint prosthesis can have several outcomes, the most feared of which is trans-femoral amputation. In order to save the limb while maintaining function, the management of these infections involves several specialists. Orthopedic surgeons are on the front line for carrying out bacteriological samples as well as for changing the material when necessary. The infectiologists coordinate this care by supervising each of the interventions by an antibiotic therapy adapted to the germs and by ensuring the occurrence of adverse events related to the treatment. Plastic surgeons intervene when the skin cover of the knee is deemed to be precarious or when there is an identified loss of substance that could affect the prognosis of the prosthesis. The main objective of our study is to evaluate the success rate of skin coverage and functional recovery for patients cured of their infection. The secondary objective is the identification of risk factors for skin coverage in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a prosthesis knee infection whose management requires skin covering plastic surgery
* Surgical procedures performed at the Croix Rousse Hospital

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a prosthesis knee infection infection whose management requires skin covering plastic surgery
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
rate of patients with prosthesis knee infection requiring skin coverage | 2011-2021
  proportion of patients with prosthesis knee infection requiring skin coverage amaong all prosthesis knee infection

SECONDARY OUTCOMES:
description of the population at risk of coverage after prosthesis knee infection | 2011-2021
  rate of failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: website of crioac lyon — https://www.crioac-lyon.fr/en/